CLINICAL TRIAL: NCT00658814
Title: A Phase II Trial of Azacitidine (NSC-102816) Plus Gemtuzumab Ozogamicin (NSC-720568) as Induction and Post-Remission Therapy in Patients of Age 60 and Older With Previously Untreated Non-M3 Acute Myeloid Leukemia
Brief Title: Azacitidine and Gemtuzumab Ozogamicin in Treating Older Patients With Previously Untreated Acute Myeloid Leukemia
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2009-00790; NCI-2009-00790 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); SWOG-S0703; CDR0000593117; S0703 (Other: SWOG); S0703 (Other: CTEP); U10CA032102 (NIH)
Record Dates: First submitted 2008-04-12; First posted 2008-04-15 (Estimated); Results first posted 2014-01-06 (Estimated); Last update posted 2025-07-28 (Actual); Status verified 2025-06

CONDITIONS: Acute Myeloid Leukemia; Adult Acute Megakaryoblastic Leukemia; Adult Acute Monoblastic Leukemia; Adult Acute Monocytic Leukemia; Adult Acute Myeloid Leukemia With Inv(16)(p13.1q22); CBFB-MYH11; Adult Acute Myeloid Leukemia With Maturation; Adult Acute Myeloid Leukemia With t(16;16)(p13.1;q22); CBFB-MYH11; Adult Acute Myeloid Leukemia With t(8;21); (q22; q22.1); RUNX1-RUNX1T1; Adult Acute Myeloid Leukemia With t(9;11)(p21.3;q23.3); MLLT3-KMT2A; Adult Acute Myeloid Leukemia Without Maturation; Adult Acute Myelomonocytic Leukemia; Adult Erythroleukemia; Adult Pure Erythroid Leukemia; Secondary Acute Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Leukemia, Megakaryoblastic, Acute; Leukemia, Monocytic, Acute; Leukemia, Myelomonocytic, Acute; Leukemia, Erythroblastic, Acute | interventions — Azacitidine; Gemtuzumab

ARMS (1):
- Treatment (azacitidine, gemtuzumab) (Experimental): See Detailed Description
  Interventions: Drug: Azacitidine; Drug: Gemtuzumab Ozogamicin

INTERVENTIONS:
Drug: Azacitidine — Given IV or SC during induction; given SC during consolidation and maintenance
  Other Names: 5 AZC; 5-AC; 5-Azacitidine; 5-Azacytidine; 5-AZC; Azacytidine; Azacytidine, 5-; Ladakamycin; Mylosar; U-18496; Vidaza
Drug: Gemtuzumab Ozogamicin — Given IV
  Other Names: Calicheamicin-Conjugated Humanized Anti-CD33 Monoclonal Antibody; CDP-771; CMA-676; gemtuzumab; hP67.6-Calicheamicin; Mylotarg; WAY-CMA-676

SUMMARY:
This phase II trial is studying the side effects of giving azacitidine together with gemtuzumab ozogamicin to see how well it works in treating older patients with previously untreated acute myeloid leukemia. Drugs used in chemotherapy, such as azacitidine, work in different ways to stop the growth of cancer cells, either by killing the cells or by stopping them from dividing. Azacitidine may also stop the growth of cancer cells by blocking some of the enzymes needed for cell growth. Monoclonal antibodies, such as gemtuzumab ozogamicin, can block cancer growth in different ways. Some block the ability of cancer cells to grow and spread. Others find cancer cells and help kill them or carry cancer-killing substances to them. Giving azacitidine together with gemtuzumab ozogamicin may kill more cancer cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To test whether outcomes of patients of age 60 or older with previously untreated non-M3 acute myeloid leukemia treated with azacitidine plus gemtuzumab ozogamicin are sufficient to warrant phase III investigation.

II. To estimate the frequency and severity of toxicities of this regimen in the good- and poor-risk groups of patients.

III. To investigate in a preliminary manner the disease-free survival of patients who achieve complete remission and receive post-remission therapy on this study.

IV. To investigate in a preliminary manner the cytogenetic response rates of patients treated with this regimen.

V. To investigate in a preliminary manner the effects of cytogenetic abnormalities, promoter and global methylation changes, and multidrug resistance on overall survival and response to azacitidine plus gemtuzumab ozogamicin therapy.

OUTLINE: Patients are stratified according to risk status (good [60-69 years of age OR Zubrod performance status [PS] 0-1] vs poor [>= 70 years of age AND Zubrod PS 2-3]).

REMISSION INDUCTION THERAPY: Patients receive azacitidine intravenously (IV) over 10-40 minutes or subcutaneously (SC) once daily (QD) on days 1-7 and gemtuzumab ozogamicin IV over 2 hours on day 8. Patients with residual leukemia (blast count >= 5%) receive a second course of induction therapy beginning between days 15-29. Patients achieving complete remission (CR) or morphologic complete remission with incomplete blood count recovery (CRi) go on to receive consolidation therapy.

CONSOLIDATION THERAPY: Patients receive one course of azacitidine and gemtuzumab ozogamicin as in induction therapy (with azacitidine given SC only).

MAINTENANCE THERAPY: Patients receive azacitidine SC on days 1-7. Treatment repeats every 28 days for 4 courses in the absence of disease progression or unacceptable toxicity. Patients undergo bone marrow biopsies for cytogenetic studies at baseline, remission, and relapse or progression (and at completion of treatment if it does not correspond to one of these time points). Marrow and blood samples are submitted to correlatives studies and submitted to Southwest Oncology Group (SWOG) acute lymphoblastic leukemia (ALL)/chronic lymphocytic leukemia (CLL)/chronic myelogenous leukemia (CML) Repository in Seattle, WA.

After completion of study therapy, patients are followed every 2 months for 2 years, every 3 months for 1 year, every 4 months for 1 year, and then every 6 months thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Morphologically confirmed diagnosis of acute myeloid leukemia (AML) with classification other than WHO acute promyelocytic leukemia (FAB M3), based on bone marrow examination performed within 14 days prior to registration; patients with World Health Organization (WHO) acute promyelocytic leukemia (FAB M3) or blastic transformation of chronic myelogenous leukemia are not eligible
* Zubrod performance status 0-3
* No known hypersensitivity to azacitidine, mannitol, hydroxyurea, orgemtuzumab ozogamicin
* No prior systemic chemotherapy for acute leukemia with the exception of hydroxyurea; administration of hydroxyurea to control high white blood cell (WBC) count prior to registration is permitted
* Patients with a history of prior myelodysplastic syndrome (MDS) are eligible according to the following criteria:

  * No prior treatment of MDS with AML induction-type chemotherapy or high-dose chemotherapy with hematopoietic stem cell support
  * Prior cytarabine allowed if dose < 100 mg/m^2/day
  * Prior hematopoietic growth factors, thalidomide, lenalidomide, arsenic trioxide, and signal transduction inhibitors for treatment of MDS allowed
  * No prior treatment with azacitidine, decitabine, or gemtuzumab ozogamicin
  * At least 30 days since prior therapy for MDS and recovered
* Bilirubin =< 2.0 x institutional upper limit of normal (IULN) within 14 days to registration, unless the elevation is believed to be due to hepatic infiltration by AML

  * Hyperbilirubinemia due primarily to elevated unconjugated hyperbilirubinemia secondary to Gilbert syndrome or hemolysis is allowed
* Serum glutamic oxaloacetic transaminase (SGOT) aspartate aminotransferase (AST) =< 2 x IULN, or serum glutamic pyruvate transaminase (SGPT) alanine aminotransferase (ALT) =< 2.0 x IULN , unless the elevation is believed to be due to hepatic infiltration by AML
* Serum creatinine =< 1.5 x IULN
* Left ventricle ejection fraction (LVEF) >= 40% by multi-gated acquisition scan (MUGA) or echocardiogram (ECHO) AND no clinical evidence of congestive heart failure within the past 56 days
* Pretreatment cytogenetics must be performed on all patients; collection of pretreatment specimens must be completed within 14 days prior to registration to S0703; specimens must be submitted to the site's preferred cytogenetics laboratory
* Patients must consent to submit specimens to the Southwest Oncology Group (SWOG) acute lymphoblastic leukemia (ALL)/chronic lymphocytic leukemia (CLL)/chronic myelogenous leukemia (CML) repository for cellular and molecular studies; collection of pretreatment blood and/or marrow specimens must be completed within 14 days prior to registration; if a marrow specimen is available, either from the diagnostic marrow or a repeat pre-registration marrow, then it must be submitted along with a peripheral blood specimen; otherwise peripheral blood alone must be submitted; residual specimens will only be banked if the patient provides separate consent; sites are required to offer patients the opportunity to participate in banking
* No central nervous system (CNS) involvement; if central nervous involvement is clinically suspected, it must be ruled out by a lumbar puncture
* Women of reproductive potential must have a pregnancy test within 28 days prior to registration; patients must not be pregnant or nursing because of the teratogenic potential of the drugs used in this study; women/men of reproductive potential must have agreed to use an effective contraceptive method
* Patients not known to be human immunodeficiency virus positive (HIV+) must be tested for HIV infection within 14 days prior to registration
* HIV-positive patients must meet the following criteria:

  * No history of acquired immunodeficiency syndrome (AIDS)-defining events
  * CD4 cells >= 500/mm^3
  * Viral load of < 50 copies HIV messenger ribonucleic acid (mRNA)/mm^3 if on cART or < 25,000 copies HIV mRNA if not on cART
  * No zidovudine or stavudine as part of cART Patients who are HIV+ and do not meet all of these criteria will not be eligible for this study
* No other prior malignancy except for a) adequately treated basal cell or squamous cell skin cancer or b) any diagnosis of malignancy made within the past 2 years earlier, of which there is no clinically evident cancer, and for which the patient has completed all chemotherapy and radiotherapy at least 6 months prior to study registration; prior treatment with AML induction-type chemotherapy is not allowed; concurrent hormonal therapy is allowed
* All patients must be informed of the investigational nature of this study and must sign and give written informed consent in accordance with institutional and federal guidelines
* At the time of patient registration, the treating institution's name and identification (ID) number must be provided to the Data Operations Center in Seattle in order to ensure that the current (within 365 days) date of institutional review board approval for this study has been entered into the data base
* Patients must have complete remission (CR) or CRi, documented by blood and marrow examinations performed within 42 days before this registration
* Following completion of induction therapy, the blood counts must recover to absolute neutrophil count (ANC) >= 1,000/mcL and platelets >= 90,000/mcL (without transfusion), and must be maintained at these levels during the 7 days prior to registration
* Patients must have serum creatinine =< 1.5 x IULN and SGOT or SGPT =< 1.5 x IULN within 28 days before registration
* Patients must have recovered to =< Grade 2 from any induction cycle non-hematologic toxicities

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 133 (Actual)
Dates: Start 2008-12-01 (Actual); Primary Completion 2013-06-01 (Actual); Study Completion 2026-03-19 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Sucha Nand, Principal Investigator — SWOG Cancer Research Network
Locations (177):
- United States (177):
  - Providence Saint Joseph Medical Center/Disney Family Cancer Center, Burbank, California
  - Stanford Cancer Institute Palo Alto, Palo Alto, California
  - University of California Davis Comprehensive Cancer Center, Sacramento, California
  - Smilow Cancer Hospital Care Center at Saint Francis, Hartford, Connecticut
  - Saint Alphonsus Cancer Care Center-Boise, Boise, Idaho
  - OSF Saint Anthony's Health Center, Alton, Illinois
  - Decatur Memorial Hospital, Decatur, Illinois
  - Heartland Cancer Research NCORP, Decatur, Illinois
  - Advocate Sherman Hospital, Elgin, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - SSM Health Good Samaritan, Mount Vernon, Illinois
  - Springfield Memorial Hospital, Springfield, Illinois
  - Franciscan Saint Francis Health-Beech Grove, Beech Grove, Indiana
  - Reid Health, Richmond, Indiana
  - Hospital District Sixth of Harper County, Anthony, Kansas
  - Cancer Center of Kansas - Chanute, Chanute, Kansas
  - Cancer Center of Kansas - Dodge City, Dodge City, Kansas
  - Cancer Center of Kansas - El Dorado, El Dorado, Kansas
  - Cancer Center of Kansas - Fort Scott, Fort Scott, Kansas
  - Cancer Center of Kansas-Independence, Independence, Kansas
  - Cancer Center of Kansas-Kingman, Kingman, Kansas
  - Lawrence Memorial Hospital, Lawrence, Kansas
  - Southwest Medical Center, Liberal, Kansas
  - Cancer Center of Kansas-Liberal, Liberal, Kansas
  - Cancer Center of Kansas - Newton, Newton, Kansas
  - Menorah Medical Center, Overland Park, Kansas
  - Saint Luke's South Hospital, Overland Park, Kansas
  - Cancer Center of Kansas - Parsons, Parsons, Kansas
  - Kansas City NCI Community Oncology Research Program, Prairie Village, Kansas
  - Cancer Center of Kansas - Pratt, Pratt, Kansas
  - Cancer Center of Kansas - Salina, Salina, Kansas
  - Salina Regional Health Center, Salina, Kansas
  - AdventHealth Shawnee Mission, Shawnee Mission, Kansas
  - Cotton O'Neil Cancer Center / Stormont Vail Health, Topeka, Kansas
  - Cancer Center of Kansas - Wellington, Wellington, Kansas
  - Associates In Womens Health, Wichita, Kansas
  - Cancer Center of Kansas-Wichita Medical Arts Tower, Wichita, Kansas
  - Ascension Via Christi Hospitals Wichita, Wichita, Kansas
  - Cancer Center of Kansas - Wichita, Wichita, Kansas
  - Wesley Medical Center, Wichita, Kansas
  - Wichita NCI Community Oncology Research Program, Wichita, Kansas
  - Cancer Center of Kansas - Winfield, Winfield, Kansas
  - University of Kentucky/Markey Cancer Center, Lexington, Kentucky
  - Hematology/Oncology Clinic PLLC, Baton Rouge, Louisiana
  - Tulane University School of Medicine, New Orleans, Louisiana
  - Michigan Cancer Research Consortium NCORP, Ann Arbor, Michigan
  - Trinity Health Saint Joseph Mercy Hospital Ann Arbor, Ann Arbor, Michigan
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Bronson Battle Creek, Battle Creek, Michigan
  - Spectrum Health Big Rapids Hospital, Big Rapids, Michigan
  - Corewell Health Dearborn Hospital, Dearborn, Michigan
  - Wayne State University/Karmanos Cancer Institute, Detroit, Michigan
  - Henry Ford Health Saint John Hospital, Detroit, Michigan
  - Hurley Medical Center, Flint, Michigan
  - Genesys Regional Medical Center-West Flint Campus, Flint, Michigan
  - Cancer Research Consortium of West Michigan NCORP, Grand Rapids, Michigan
  - Corewell Health Grand Rapids Hospitals - Butterworth Hospital, Grand Rapids, Michigan
  - Trinity Health Grand Rapids Hospital, Grand Rapids, Michigan
  - Allegiance Health, Jackson, Michigan
  - University of Michigan Health - Sparrow Lansing, Lansing, Michigan
  - Trinity Health Saint Mary Mercy Livonia Hospital, Livonia, Michigan
  - Trinity Health Muskegon Hospital, Muskegon, Michigan
  - Trinity Health Saint Joseph Mercy Oakland Hospital, Pontiac, Michigan
  - Lake Huron Medical Center, Port Huron, Michigan
  - MyMichigan Medical Center Saginaw, Saginaw, Michigan
  - Henry Ford Health Providence Southfield Hospital, Southfield, Michigan
  - Munson Medical Center, Traverse City, Michigan
  - Henry Ford Health Warren Hospital, Warren, Michigan
  - University of Michigan Health - West, Wyoming, Michigan
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Southeast Missouri Hospital, Cape Girardeau, Missouri
  - Saint Francis Medical Center, Cape Girardeau, Missouri
  - University Health Truman Medical Center, Kansas City, Missouri
  - Saint Luke's Hospital of Kansas City, Kansas City, Missouri
  - Saint Joseph Health Center, Kansas City, Missouri
  - North Kansas City Hospital, Kansas City, Missouri
  - Heartland Hematology and Oncology Associates Incorporated, Kansas City, Missouri
  - Research Medical Center, Kansas City, Missouri
  - Saint Luke's East - Lee's Summit, Lee's Summit, Missouri
  - Liberty Hospital, Liberty, Missouri
  - Heartland Regional Medical Center, Saint Joseph, Missouri
  - Mercy Infusion Center - Chippewa, St Louis, Missouri
  - Mercy Hospital Saint Louis, St Louis, Missouri
  - Saint Louis-Cape Girardeau CCOP, St Louis, Missouri
  - Billings Clinic Cancer Center, Billings, Montana
  - Northern Rockies Radiation Oncology Center, Billings, Montana
  - Saint Vincent Healthcare, Billings, Montana
  - Montana Cancer Consortium NCORP, Billings, Montana
  - Saint Vincent Frontier Cancer Center, Billings, Montana
  - Bozeman Health Deaconess Hospital, Bozeman, Montana
  - Saint James Community Hospital and Cancer Treatment Center, Butte, Montana
  - Benefis Sletten Cancer Institute, Great Falls, Montana
  - Berdeaux, Donald MD (UIA Investigator), Great Falls, Montana
  - Great Falls Clinic, Great Falls, Montana
  - Northern Montana Hospital, Havre, Montana
  - Saint Peter's Community Hospital, Helena, Montana
  - Glacier Oncology PLLC, Kalispell, Montana
  - Kalispell Medical Oncology, Kalispell, Montana
  - Logan Health Medical Center, Kalispell, Montana
  - Montana Cancer Specialists, Missoula, Montana
  - Saint Patrick Hospital - Community Hospital, Missoula, Montana
  - Community Medical Center, Missoula, Montana
  - Guardian Oncology and Center for Wellness, Missoula, Montana
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
  - University of Rochester, Rochester, New York
  - Novant Health Presbyterian Medical Center, Charlotte, North Carolina
  - Wayne Memorial Hospital, Goldsboro, North Carolina
  - Margaret R Pardee Memorial Hospital, Hendersonville, North Carolina
  - Rutherford Hospital, Rutherfordton, North Carolina
  - Southeast Clinical Oncology Research Consortium NCORP, Winston-Salem, North Carolina
  - Cleveland Clinic Akron General, Akron, Ohio
  - Mary Rutan Hospital, Bellefontaine, Ohio
  - Adena Regional Medical Center, Chillicothe, Ohio
  - University of Cincinnati Cancer Center-UC Medical Center, Cincinnati, Ohio
  - Riverside Methodist Hospital, Columbus, Ohio
  - Columbus NCI Community Oncology Research Program, Columbus, Ohio
  - Grant Medical Center, Columbus, Ohio
  - Mount Carmel Health Center West, Columbus, Ohio
  - Doctors Hospital, Columbus, Ohio
  - Grandview Hospital, Dayton, Ohio
  - Good Samaritan Hospital - Dayton, Dayton, Ohio
  - Miami Valley Hospital, Dayton, Ohio
  - Miami Valley Hospital North, Dayton, Ohio
  - Dayton NCI Community Oncology Research Program, Dayton, Ohio
  - Grady Memorial Hospital, Delaware, Ohio
  - Blanchard Valley Hospital, Findlay, Ohio
  - Atrium Medical Center-Middletown Regional Hospital, Franklin, Ohio
  - Wayne Hospital, Greenville, Ohio
  - Kettering Medical Center, Kettering, Ohio
  - Fairfield Medical Center, Lancaster, Ohio
  - Marietta Memorial Hospital, Marietta, Ohio
  - Knox Community Hospital, Mount Vernon, Ohio
  - Licking Memorial Hospital, Newark, Ohio
  - Southern Ohio Medical Center, Portsmouth, Ohio
  - Springfield Regional Medical Center, Springfield, Ohio
  - Upper Valley Medical Center, Troy, Ohio
  - Saint Ann's Hospital, Westerville, Ohio
  - Clinton Memorial Hospital/Foster J Boyd Regional Cancer Center, Wilmington, Ohio
  - Greene Memorial Hospital, Xenia, Ohio
  - Genesis Healthcare System Cancer Care Center, Zanesville, Ohio
  - Clackamas Radiation Oncology Center, Clackamas, Oregon
  - Legacy Mount Hood Medical Center, Gresham, Oregon
  - Providence Milwaukie Hospital, Milwaukie, Oregon
  - Providence Newberg Medical Center, Newberg, Oregon
  - Providence Willamette Falls Medical Center, Oregon City, Oregon
  - Legacy Good Samaritan Hospital and Medical Center, Portland, Oregon
  - Providence Portland Medical Center, Portland, Oregon
  - Adventist Medical Center, Portland, Oregon
  - Providence Saint Vincent Medical Center, Portland, Oregon
  - Legacy Emanuel Hospital and Health Center, Portland, Oregon
  - Salem Hospital, Salem, Oregon
  - Legacy Meridian Park Hospital, Tualatin, Oregon
  - AnMed Health Hospital, Anderson, South Carolina
  - Medical University of South Carolina, Charleston, South Carolina
  - Spartanburg Medical Center, Spartanburg, South Carolina
  - The Don and Sybil Harrington Cancer Center, Amarillo, Texas
  - Cancer Care Center at Island Hospital, Anacortes, Washington
  - PeaceHealth Saint Joseph Medical Center, Bellingham, Washington
  - Highline Medical Center-Main Campus, Burien, Washington
  - Swedish Cancer Institute-Issaquah, Issaquah, Washington
  - Kadlec Clinic Hematology and Oncology, Kennewick, Washington
  - Skagit Valley Hospital, Mount Vernon, Washington
  - Harrison HealthPartners Hematology and Oncology-Poulsbo, Poulsbo, Washington
  - Harborview Medical Center, Seattle, Washington
  - Minor and James Medical PLLC, Seattle, Washington
  - Fred Hutchinson Cancer Center, Seattle, Washington
  - Kaiser Permanente Washington, Seattle, Washington
  - Swedish Medical Center-First Hill, Seattle, Washington
  - University of Washington Medical Center - Montlake, Seattle, Washington
  - PeaceHealth United General Medical Center, Sedro-Woolley, Washington
  - Saint Michael Cancer Center, Silverdale, Washington
  - Cancer Care Northwest - Spokane South, Spokane, Washington
  - Evergreen Hematology and Oncology PS, Spokane, Washington
  - PeaceHealth Southwest Medical Center, Vancouver, Washington
  - Wenatchee Valley Hospital and Clinics, Wenatchee, Washington
  - Rocky Mountain Oncology, Casper, Wyoming
  - Welch Cancer Center, Sheridan, Wyoming

REFERENCES:
- [Derived] Nand S, Othus M, Godwin JE, Willman CL, Norwood TH, Howard DS, Coutre SE, Erba HP, Appelbaum FR. A phase 2 trial of azacitidine and gemtuzumab ozogamicin therapy in older patients with acute myeloid leukemia. Blood. 2013 Nov 14;122(20):3432-9. doi: 10.1182/blood-2013-06-506592. Epub 2013 Oct 3. PMID 24092933

RESULTS

PARTICIPANT FLOW:
Groups:
- Good Risk Patients: Azacitidine Plus Gemtuzumab Ozogamicin: Good risk patients defined as those aged 60-69 or those with performance status of Zubrod 0-1.
  Remission Induction: Azacitidine intravenously (IV) over 10-40 minutes or subcutaneously (SC) once daily on days 1-7 and gemtuzumab ozogamicin IV over 2 hours on day 8. (1 cycle = 14 days)
  Patients achieving complete remission (CR) or morphologic complete remission with incomplete blood count recovery (CRi) go on to receive consolidation therapy.
  Consolidation: Azacitidine subcutaneously (SC) once daily on days 1-7 and gemtuzumab ozogamicin IV over 2 hours on day 8.
  Patients in continued remission may go on to receive maintenance therapy.
  Maintenance: Azacitidine subcutaneously on days 1-7 (1 cycle = 28 days)
- Poor Risk Patients: Azacitidine Plus Gemtuzumab Ozogamicin: Poor risk patients defined as those who were at least 70 years old and had a performance status of 2 or 3.
  Remission Induction: Azacitidine intravenously (IV) over 10-40 minutes or subcutaneously (SC) once daily on days 1-7 and gemtuzumab ozogamicin IV over 2 hours on day 8. (1 cycle = 14 days)
  Patients achieving complete remission (CR) or morphologic complete remission with incomplete blood count recovery (CRi) go on to receive consolidation therapy.
  Consolidation: Azacitidine subcutaneously (SC) once daily on days 1-7 and gemtuzumab ozogamicin IV over 2 hours on day 8.
  Patients in continued remission may go on to receive maintenance therapy.
  Maintenance: Azacitidine subcutaneously on days 1-7 (1 cycle = 28 days)
Period: Remission Induction Chemotherapy
Arm/Group | Good Risk Patients: Azacitidine Plus Gemtuzumab Ozogamicin | Poor Risk Patients: Azacitidine Plus Gemtuzumab Ozogamicin
Started | 83 | 59
Eligible | 82 | 57
Eligible and Began Protocol Therapy | 79 | 54
Completed | 75 | 41
Not Completed | 8 | 18
Not completed — Adverse Event | 1 | 3
Not completed — Withdrawal by Subject | 3 | 4
Not completed — Progression/Relapse | 0 | 1
Not completed — Death | 1 | 4
Not completed — Not protocol specified | 2 | 4
Not completed — Not eligible | 1 | 2
Period: Consolidation Therapy
Arm/Group | Good Risk Patients: Azacitidine Plus Gemtuzumab Ozogamicin | Poor Risk Patients: Azacitidine Plus Gemtuzumab Ozogamicin
Started | 24 | 13
Eligible | 22 | 11
Completed | 22 | 10
Not Completed | 2 | 3
Not completed — Not protocol specified | 0 | 1
Not completed — Not eligible | 2 | 2
Period: Maintenance Therapy
Arm/Group | Good Risk Patients: Azacitidine Plus Gemtuzumab Ozogamicin | Poor Risk Patients: Azacitidine Plus Gemtuzumab Ozogamicin
Started | 20 | 8
Eligible | 19 | 8
Completed | 17 | 7
Not Completed | 3 | 1
Not completed — Adverse Event | 1 | 1
Not completed — Not protocol specified | 1 | 0
Not completed — Not eligible | 1 | 0

BASELINE CHARACTERISTICS:
Population: Eligible patients who began protocol therapy
Groups:
- Good Risk Patients: Azacitidine Plus Gemtuzumab Ozogamicin: Good risk patients defined as those aged 60-69 or those with performance status of Zubrod 0-1.
  Remission Induction: Azacitidine intravenously (IV) over 10-40 minutes or subcutaneously (SC) once daily on days 1-7 and gemtuzumab ozogamicin IV over 2 hours on day 8. (1 cycle = 14 days)
  Consolidation: Azacitidine subcutaneously (SC) once daily on days 1-7 and gemtuzumab ozogamicin IV over 2 hours on day 8.
  Maintenance: Azacitidine subcutaneously on days 1-7 (1 cycle = 28 days)
- Poor Risk Patients: Azacitidine Plus Gemtuzumab Ozogamicin: Poor risk patients defined as those who were at least 70 years old and had a performance status of 2 or 3.
  Remission Induction: Azacitidine intravenously (IV) over 10-40 minutes or subcutaneously (SC) once daily on days 1-7 and gemtuzumab ozogamicin IV over 2 hours on day 8. (1 cycle = 14 days)
  Consolidation: Azacitidine subcutaneously (SC) once daily on days 1-7 and gemtuzumab ozogamicin IV over 2 hours on day 8.
  Maintenance: Azacitidine subcutaneously on days 1-7 (1 cycle = 28 days)
- Total: Total of all reporting groups
Arm/Group | Good Risk Patients: Azacitidine Plus Gemtuzumab Ozogamicin | Poor Risk Patients: Azacitidine Plus Gemtuzumab Ozogamicin | Total
Number analyzed (Participants) | 79 | 54 | 133
Age, Continuous [Median (Full Range); unit: years] | 71.2 [60.5 to 88.7] | 76 [70.3 to 87] | 73.4 [60.5 to 88.7]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30 | 21 | 51
  Male | 49 | 33 | 82
Race/Ethnicity, Customized [Number; unit: participants]
  Asian | 1 | 0 | 1
  Black or African American | 1 | 4 | 5
  White | 77 | 50 | 127
Hispanic [Number; unit: participants]
  Yes | 3 | 1 | 4
  No | 64 | 50 | 114
  Unknown | 12 | 3 | 15

OUTCOME MEASURES:

1. Secondary Outcome: Number of Patients With Grade 3 Through 5 Adverse Events That Are Related to Study Drug
Description: Only adverse events that are possibly, probably or definitely related to study drug are reported.
Time Frame: Up to 5 years
Population: Eligible patients who received any treatment were included in the adverse event summaries. Any CTCAE 3.0 event of Grade 3 (severe), Grade 4 (life threatening) or Grade 5 (fatal) which were deemed to be related to protocol treatment are included.
Measure: Number; unit: Participants
Groups:
- Remission Induction Chemotherapy: Azacitidine intravenously (IV) over 10-40 minutes or subcutaneously (SC) once daily on days 1-7 and gemtuzumab ozogamicin IV over 2 hours on day 8. (1 cycle = 14 days)
- Consolidation Therapy: Azacitidine subcutaneously (SC) once daily on days 1-7 and gemtuzumab ozogamicin IV over 2 hours on day 8.
- Maintenance Therapy: Azacitidine subcutaneously on days 1-7 (1 cycle = 28 days)
Arm/Group | Remission Induction Chemotherapy | Consolidation Therapy | Maintenance Therapy
Number analyzed (Participants) | 133 | 32 | 27
Participants
  ALT, SGPT (serum glutamic pyruvic transaminase) | 5 | 0 | 0
  AST, SGOT | 4 | 0 | 0
  Adult respiratory distress syndrome (ARDS) | 1 | 0 | 0
  Albumin, serum-low (hypoalbuminemia) | 5 | 1 | 0
  Anorexia | 5 | 1 | 0
  Bilirubin (hyperbilirubinemia) | 3 | 0 | 0
  Calcium, serum-low (hypocalcemia) | 6 | 0 | 0
  Carbon monoxide diffusion capacity (DL(co)) | 1 | 0 | 0
  Cardiac Arrhythmia-Atrial fibrilation | 1 | 0 | 0
  Cardiac General-cardiopulmonary disease | 1 | 0 | 0
  Cardiac General-Chest Pain | 1 | 0 | 0
  Cardiac troponin I (cTnI) | 1 | 0 | 0
  Cardiac-ischemia/infarction | 1 | 0 | 0
  Conduction abnormality NOS | 1 | 0 | 0
  Confusion | 1 | 0 | 0
  Constipation | 2 | 0 | 0
  Cytokine release syndrome/acute infusion reaction | 1 | 0 | 0
  Death - Disease progression NOS | 1 | 0 | 0
  Death - Multi-organ failure | 2 | 0 | 0
  Death not associated with CTCAE term - Death NOS | 1 | 0 | 0
  Dehydration | 1 | 0 | 0
  Diarrhea | 2 | 0 | 0
  Dyspnea (shortness of breath) | 5 | 1 | 2
  Edema: limb | 1 | 0 | 0
  Fatigue (asthenia, lethargy, malaise) | 18 | 1 | 1
  Febrile neutropenia | 50 | 0 | 0
  Glucose, serum-high (hyperglycemia) | 10 | 3 | 2
  Hemoglobin | 73 | 1 | 1
  Hemorrhage, CNS | 1 | 0 | 0
  Hemorrhage, GI - Stomach | 1 | 0 | 0
  Hemorrhage, GI - Upper GI NOS | 1 | 0 | 0
  Hemorrhage/Bleeding-platelets and red blood cells | 1 | 0 | 0
  Hepatobiliary/Pancreas-venoocclusive disease | 1 | 0 | 0
  Hypertension | 1 | 0 | 0
  Hypotension | 2 | 0 | 0
  Hypoxia | 4 | 0 | 0
  Inf (clin/microbio) w/Gr 3-4 neuts - Blood | 16 | 0 | 1
  Inf (clin/microbio) w/Gr 3-4 neuts - Catheter-rel | 2 | 1 | 0
  Inf (clin/microbio) w/Gr 3-4 neuts - Colon | 1 | 0 | 0
  Inf (clin/microbio) w/Gr 3-4 neuts - Conjunctiva | 1 | 0 | 0
  Inf (clin/microbio) w/Gr 3-4 neuts - Dental-tooth | 3 | 0 | 0
  Inf (clin/microbio) w/Gr 3-4 neuts - Kidney | 1 | 0 | 0
  Inf (clin/microbio) w/Gr 3-4 neuts - Lung | 8 | 0 | 0
  Inf (clin/microbio) w/Gr 3-4 neuts - Oral cav-gums | 1 | 0 | 0
  Inf (clin/microbio) w/Gr 3-4 neuts - Sinus | 2 | 0 | 0
  Inf (clin/microbio) w/Gr 3-4 neuts - Skin | 6 | 0 | 0
  Inf (clin/microbio) w/Gr 3-4 neuts - UTI | 3 | 0 | 0
  Inf w/normal ANC or Gr 1-2 neutrophils - Blood | 2 | 1 | 0
  Inf w/normal ANC or Gr 1-2 neutrophils - Lung | 0 | 0 | 1
  Inf w/normal ANC or Gr 1-2 neutrophils - Skin | 1 | 0 | 0
  Infection with unknown ANC - Blood | 1 | 0 | 0
  Infection with unknown ANC - Lung (pneumonia) | 1 | 0 | 0
  Infection with unknown ANC - Skin (cellulitis) | 1 | 0 | 0
  Infection-Aspirgillosis | 1 | 0 | 0
  Infection-bacteremia | 1 | 0 | 0
  Left ventricular systolic dysfunction | 1 | 0 | 0
  Leukocytes (total WBC) | 80 | 18 | 6
  Liver dysfunction/failure (clinical) | 0 | 1 | 0
  Lymphopenia | 23 | 0 | 1
  Mood alteration - depression | 2 | 0 | 0
  Mucositis/stomatitis (functional/symp) - Oral cav | 1 | 0 | 0
  Muscle weakness, not d/t neuropathy - body/general | 4 | 0 | 0
  Neutrophils/granulocytes (ANC/AGC) | 85 | 21 | 10
  Pain - Cardiac/heart | 2 | 0 | 0
  Petechiae/purpura (hemorrhage into skin or mucosa) | 1 | 0 | 0
  Phosphate, serum-low (hypophosphatemia) | 4 | 0 | 0
  Platelets | 85 | 12 | 3
  Pleural effusion (non-malignant) | 1 | 0 | 0
  Pneumonitis/pulmonary infiltrates | 1 | 0 | 0
  Potassium, serum-low (hypokalemia) | 5 | 0 | 0
  Pulmonary/Upper Respiratory-pulmonary edema | 2 | 0 | 0
  Rash/desquamation | 1 | 0 | 0
  SVT and nodal arrhythmia - Atrial fibrillation | 2 | 0 | 0
  SVT and nodal arrhythmia - SVT tachycardia | 1 | 0 | 0
  Sodium, serum-low (hyponatremia) | 5 | 0 | 0
  Sudden death | 1 | 0 | 0
  Thrombosis/thrombus/embolism | 2 | 0 | 0

2. Primary Outcome: Complete Response
Description: Morphologic complete remission (CR): ANC >=1,000/mcL, platelet count >=100,000/mcL, <5% bone marrow blasts, no Auer rods, no evidence of extramedullary disease. Morphologic complete remission with incomplete blood count recovery (CRi): Same as CR but ANC may be <1,000/mcL and/or platelet count <100,000/mcL.
Time Frame: Up to 60 days
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Good Risk Patients: Azacitidine Plus Gemtuzumab Ozogamicin | Poor Risk Patients: Azacitidine Plus Gemtuzumab Ozogamicin
Number analyzed (Participants) | 79 | 54
percentage of participants | 44 [33 to 56] | 35 [23 to 49]

3. Primary Outcome: 30-Day Survival
Description: Patients surviving more than 30 days after study registration
Time Frame: 30 days
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Good Risk Patients: Azacitidine Plus Gemtuzumab Ozogamicin | Poor Risk Patients: Azacitidine Plus Gemtuzumab Ozogamicin
Number analyzed (Participants) | 79 | 54
percentage of participants | 92 [84 to 97] | 87 [75 to 95]

4. Secondary Outcome: Relapse-free Survival
Description: Relapse-free survival (RFS) is defined for all patients who achieve CR or CRi. RFS is measured from the date CR or CRi is first achieved until relapse or death form any cause, with observation censored on the date of last contact for patients last known to be alive without report of relapse. Relapse from CR/CRi is defined as reappearance of leukemic blasts in the peripheral blood; or > 5% blasts in the bone marrow not attributable to another cause; or appearance or reappearance of extramedullary disease.
Time Frame: Up to 5 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Good Risk Patients: Azacitidine Plus Gemtuzumab Ozogamicin | Poor Risk Patients: Azacitidine Plus Gemtuzumab Ozogamicin
Number analyzed (Participants) | 35 | 19
months | 8 [5 to 13] | 7 [6 to 12]

ADVERSE EVENTS:
Time Frame: Up to 5 years
Arm/Group | Remission Induction Chemotherapy | Consolidation Therapy | Maintenance Therapy
Serious Adverse Events (participants affected / at risk) | 55/133 | 1/32 | 3/27
Other Adverse Events (participants affected / at risk) | 130/133 | 32/32 | 26/27
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Remission Induction Chemotherapy (N=133) | Consolidation Therapy (N=32) | Maintenance Therapy (N=27)
Febrile neutropenia (Blood and lymphatic system disorders) | 10 | 0 | 0
Hemoglobin (Blood and lymphatic system disorders) | 4 | 0 | 0
Cardiac-ischemia/infarction (Cardiac disorders) | 2 | 0 | 0
Conduction abnormality NOS (Cardiac disorders) | 1 | 0 | 0
Left ventricular systolic dysfunction (Cardiac disorders) | 2 | 0 | 0
Pain - Cardiac/heart (Cardiac disorders) | 1 | 0 | 0
SVT and nodal arrhythmia - Atrial fibrillation (Cardiac disorders) | 3 | 0 | 0
SVT and nodal arrhythmia - SVT tachycardia (Cardiac disorders) | 1 | 0 | 0
SVT and nodal arrhythmia - Sinus tachycardia (Cardiac disorders) | 1 | 0 | 0
Ventricular arrhythmia - Ventricular fibrillation (Cardiac disorders) | 1 | 0 | 0
Colitis (Gastrointestinal disorders) | 1 | 0 | 0
Hemorrhage, GI - Stomach (Gastrointestinal disorders) | 1 | 0 | 0
Hemorrhage, GI - Upper GI NOS (Gastrointestinal disorders) | 1 | 0 | 0
Ileus, GI (functional obstruction of bowel) (Gastrointestinal disorders) | 1 | 0 | 0
Obstruction, GI - Small bowel NOS (Gastrointestinal disorders) | 1 | 0 | 0
Death - Multi-organ failure (General disorders) | 2 | 0 | 0
Death not associated with CTCAE term - Death NOS (General disorders) | 2 | 0 | 0
Fatigue (asthenia, lethargy, malaise) (General disorders) | 1 | 0 | 0
Sudden death (General disorders) | 2 | 0 | 0
Liver dysfunction/failure (clinical) (Hepatobiliary disorders) | 0 | 1 | 0
Cytokine release syndrome/acute infusion reaction (Immune system disorders) | 1 | 0 | 0
Inf (clin/microbio) w/Gr 3-4 neuts - Blood (Infections and infestations) | 7 | 0 | 0
Inf (clin/microbio) w/Gr 3-4 neuts - Catheter-rel (Infections and infestations) | 1 | 1 | 0
Inf (clin/microbio) w/Gr 3-4 neuts - Dental-tooth (Infections and infestations) | 1 | 0 | 0
Inf (clin/microbio) w/Gr 3-4 neuts - Lung (Infections and infestations) | 7 | 0 | 0
Inf (clin/microbio) w/Gr 3-4 neuts - Sinus (Infections and infestations) | 2 | 0 | 0
Inf (clin/microbio) w/Gr 3-4 neuts - Skin (Infections and infestations) | 2 | 0 | 0
Inf (clin/microbio) w/Gr 3-4 neuts - UTI (Infections and infestations) | 1 | 0 | 0
Inf w/normal ANC or Gr 1-2 neutrophils - Blood (Infections and infestations) | 3 | 0 | 0
Inf w/normal ANC or Gr 1-2 neutrophils - Lung (Infections and infestations) | 0 | 0 | 1
Infection with unknown ANC - Blood (Infections and infestations) | 2 | 0 | 0
Infection with unknown ANC - Lung (pneumonia) (Infections and infestations) | 1 | 0 | 0
Infection-Other (Specify):bacteremia (Infections and infestations) | 1 | 0 | 0
Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Hemorrhage/bleeding w/surgery, intra- or post-op (Injury, poisoning and procedural complications) | 1 | 0 | 0
ALT, SGPT (serum glutamic pyruvic transaminase) (Investigations) | 2 | 0 | 0
AST, SGOT (Investigations) | 2 | 0 | 0
Bilirubin (hyperbilirubinemia) (Investigations) | 2 | 0 | 0
Carbon monoxide diffusion capacity (DL(co)) (Investigations) | 1 | 0 | 0
Cardiac troponin I (cTnI) (Investigations) | 2 | 0 | 0
Creatinine (Investigations) | 2 | 0 | 0
Leukocytes (total WBC) (Investigations) | 1 | 0 | 0
Neutrophils/granulocytes (ANC/AGC) (Investigations) | 3 | 0 | 0
Platelets (Investigations) | 1 | 0 | 0
Acidosis (metabolic or respiratory) (Metabolism and nutrition disorders) | 1 | 0 | 0
Albumin, serum-low (hypoalbuminemia) (Metabolism and nutrition disorders) | 1 | 0 | 0
Calcium, serum-low (hypocalcemia) (Metabolism and nutrition disorders) | 2 | 0 | 0
Glucose, serum-high (hyperglycemia) (Metabolism and nutrition disorders) | 2 | 0 | 1
Magnesium, serum-low (hypomagnesemia) (Metabolism and nutrition disorders) | 1 | 0 | 0
Phosphate, serum-low (hypophosphatemia) (Metabolism and nutrition disorders) | 1 | 0 | 0
Potassium, serum-high (hyperkalemia) (Metabolism and nutrition disorders) | 1 | 0 | 0
Tumor lysis syndrome (Metabolism and nutrition disorders) | 1 | 0 | 0
Muscle weakness, not d/t neuropathy - body/general (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Pain - Back (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Death - Disease progression NOS (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 12 | 0 | 0
Myelodysplasia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
CNS cerebrovascular ischemia (Nervous system disorders) | 1 | 0 | 0
Encephalopathy (Nervous system disorders) | 1 | 0 | 0
Hemorrhage, CNS (Nervous system disorders) | 3 | 0 | 0
Neurology-Other (Nervous system disorders) | 1 | 0 | 0
Confusion (Psychiatric disorders) | 2 | 0 | 0
Mood alteration - depression (Psychiatric disorders) | 1 | 0 | 0
Proteinuria (Renal and urinary disorders) | 1 | 0 | 0
Renal failure (Renal and urinary disorders) | 1 | 0 | 1
Carbon monoxide diffusion capacity (DL(co)) (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 5 | 0 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 4 | 0 | 0
Pleural effusion (non-malignant) (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pneumonitis/pulmonary infiltrates (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0
Pulmonary/Upper Respiratory-Other (Specify):Pulmonary Edema (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0
Pulmonary/Upper Respiratory-Other (Specify):Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Hypertension (Vascular disorders) | 1 | 0 | 0
Hypotension (Vascular disorders) | 6 | 0 | 0
Thrombosis/thrombus/embolism (Vascular disorders) | 3 | 0 | 0
Vascular-Other (Specify):pariatal to occiptal lobe (Vascular disorders) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Remission Induction Chemotherapy (N=133) | Consolidation Therapy (N=32) | Maintenance Therapy (N=27)
Febrile neutropenia (Blood and lymphatic system disorders) | 49 | 1 | 0
Hemoglobin (Blood and lymphatic system disorders) | 98 | 20 | 15
Watery eye (epiphora, tearing) (Eye disorders) | 0 | 3 | 0
Constipation (Gastrointestinal disorders) | 47 | 6 | 10
Diarrhea (Gastrointestinal disorders) | 35 | 1 | 7
Heartburn/dyspepsia (Gastrointestinal disorders) | 8 | 1 | 1
Hemorrhoids (Gastrointestinal disorders) | 8 | 0 | 1
Mucositis/stomatitis (clinical exam) - Oral cavity (Gastrointestinal disorders) | 12 | 1 | 1
Mucositis/stomatitis (functional/symp) - Oral cav (Gastrointestinal disorders) | 8 | 1 | 0
Nausea (Gastrointestinal disorders) | 56 | 5 | 5
Pain - Abdomen NOS (Gastrointestinal disorders) | 14 | 3 | 2
Vomiting (Gastrointestinal disorders) | 27 | 0 | 2
Edema: limb (General disorders) | 30 | 3 | 3
Fatigue (asthenia, lethargy, malaise) (General disorders) | 81 | 15 | 11
Fever in absence of neutropenia, ANC lt1.0x10e9/L (General disorders) | 14 | 0 | 1
Injection site reaction/extravasation changes (General disorders) | 9 | 5 | 9
Pain - Chest/thorax NOS (General disorders) | 7 | 1 | 1
Rigors/chills (General disorders) | 21 | 2 | 1
Inf (clin/microbio) w/Gr 3-4 neuts - Blood (Infections and infestations) | 15 | 1 | 1
Inf (clin/microbio) w/Gr 3-4 neuts - Skin (Infections and infestations) | 9 | 0 | 0
Inf w/normal ANC or Gr 1-2 neutrophils - Skin (Infections and infestations) | 1 | 1 | 2
ALT, SGPT (serum glutamic pyruvic transaminase) (Investigations) | 30 | 5 | 3
AST, SGOT (Investigations) | 35 | 10 | 6
Alkaline phosphatase (Investigations) | 22 | 4 | 4
Bilirubin (hyperbilirubinemia) (Investigations) | 18 | 3 | 5
Creatinine (Investigations) | 31 | 6 | 7
Leukocytes (total WBC) (Investigations) | 87 | 23 | 16
Lymphopenia (Investigations) | 40 | 4 | 1
Neutrophils/granulocytes (ANC/AGC) (Investigations) | 91 | 23 | 14
Platelets (Investigations) | 100 | 25 | 11
Weight loss (Investigations) | 13 | 3 | 3
Albumin, serum-low (hypoalbuminemia) (Metabolism and nutrition disorders) | 63 | 13 | 9
Anorexia (Metabolism and nutrition disorders) | 45 | 5 | 5
Calcium, serum-high (hypercalcemia) (Metabolism and nutrition disorders) | 3 | 3 | 3
Calcium, serum-low (hypocalcemia) (Metabolism and nutrition disorders) | 45 | 4 | 3
Glucose, serum-high (hyperglycemia) (Metabolism and nutrition disorders) | 69 | 18 | 19
Glucose, serum-low (hypoglycemia) (Metabolism and nutrition disorders) | 7 | 2 | 3
Magnesium, serum-high (hypermagnesemia) (Metabolism and nutrition disorders) | 11 | 0 | 0
Magnesium, serum-low (hypomagnesemia) (Metabolism and nutrition disorders) | 9 | 4 | 2
Phosphate, serum-low (hypophosphatemia) (Metabolism and nutrition disorders) | 19 | 1 | 0
Potassium, serum-high (hyperkalemia) (Metabolism and nutrition disorders) | 7 | 0 | 1
Potassium, serum-low (hypokalemia) (Metabolism and nutrition disorders) | 33 | 3 | 3
Sodium, serum-low (hyponatremia) (Metabolism and nutrition disorders) | 58 | 6 | 5
Muscle weakness, not d/t neuropathy - Extrem-lower (Musculoskeletal and connective tissue disorders) | 2 | 3 | 2
Muscle weakness, not d/t neuropathy - body/general (Musculoskeletal and connective tissue disorders) | 20 | 2 | 2
Pain - Back (Musculoskeletal and connective tissue disorders) | 6 | 3 | 4
Pain - Extremity-limb (Musculoskeletal and connective tissue disorders) | 8 | 3 | 5
Pain - Joint (Musculoskeletal and connective tissue disorders) | 6 | 2 | 4
Dizziness (Nervous system disorders) | 16 | 0 | 4
Neuropathy: sensory (Nervous system disorders) | 2 | 0 | 2
Pain - Head/headache (Nervous system disorders) | 14 | 0 | 1
Taste alteration (dysgeusia) (Nervous system disorders) | 9 | 0 | 2
Confusion (Psychiatric disorders) | 9 | 1 | 0
Insomnia (Psychiatric disorders) | 16 | 5 | 2
Mood alteration - anxiety (Psychiatric disorders) | 12 | 0 | 0
Mood alteration - depression (Psychiatric disorders) | 12 | 1 | 3
Glomerular filtration rate (Renal and urinary disorders) | 6 | 2 | 1
Urinary frequency/urgency (Renal and urinary disorders) | 8 | 0 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 26 | 0 | 3
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 33 | 1 | 2
Hemorrhage, pulmonary/upper respiratory - Nose (Respiratory, thoracic and mediastinal disorders) | 12 | 0 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 10 | 0 | 0
Pleural effusion (non-malignant) (Respiratory, thoracic and mediastinal disorders) | 9 | 0 | 0
Hair loss/Alopecia (scalp or body) (Skin and subcutaneous tissue disorders) | 1 | 2 | 3
Nail changes (Skin and subcutaneous tissue disorders) | 0 | 1 | 2
Petechiae/purpura (hemorrhage into skin or mucosa) (Skin and subcutaneous tissue disorders) | 16 | 1 | 0
Pruritus/itching (Skin and subcutaneous tissue disorders) | 8 | 0 | 3
Rash/desquamation (Skin and subcutaneous tissue disorders) | 29 | 3 | 3
Rash: erythema multiforme (Skin and subcutaneous tissue disorders) | 0 | 0 | 2
Sweating (diaphoresis) (Skin and subcutaneous tissue disorders) | 12 | 2 | 1
Hypotension (Vascular disorders) | 11 | 0 | 1
Metabolic/Laboratory - elevated blood urea nitrogen (Metabolism and nutrition disorders) | 11 | 1 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less